CLINICAL TRIAL: NCT07111962
Title: Effectiveness of NOA OATMAD
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Orthoapnea (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pro00154170
Record Dates: First submitted 2025-07-07; First posted 2025-08-08 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; oral appliance therapy; mandibular advancement device
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is looking at how well the OrthoApnea NOA appliance, a special custom-made mouthpiece, helps treat people with obstructive sleep apnea (OSA). OSA is a common sleep problem where a person's breathing starts and stops many times during the night. Some people find it hard to use the usual treatment, called a continuous positive airway pressure (CPAP) machine, so this mouthpiece might be an easier and more comfortable option. The study is also checking if a small tool called the Morning Aligner, worn briefly in the morning, can help move the jaw back to its normal position. This might help people feel better and reduce side effects.

The study will last for three years. During this time, researchers will watch how people do while using the OrthoApnea NOA and compare their results to those of other people who used different types of plastic mouthpieces. The main goal is to see if the NOA can cut the number of times a person stops breathing during sleep by at least half. They hope to reduce it to fewer than 5 times an hour, which is close to normal. They will also check other things like how much oxygen people get while sleeping, their weight, how sleepy they feel during the day, how comfortable the mouthpiece is, how long it lasts, and how often people keep using it.

Instead of picking who gets which mouthpiece at random, this study uses a different method. It compares new patients using the NOA to past patients who used other mouthpieces. This is more like what happens in real life at clinics. By studying both new and past data, the researchers hope to better understand how the NOA works over time and how it compares to other options. This information will help dentists, sleep doctors, and patients choose the best way to treat sleep apnea using mouthpieces.

DETAILED DESCRIPTION:
Research Proposal: Evaluating the Effectiveness of the OrthoApnea NOA Dental Appliance in Treating Obstructive Sleep Apnea (OSA)

1. Purpose of the Study This study will evaluate how effective the OrthoApnea NOA dental appliance is at treating patients with mild, moderate, and severe obstructive sleep apnea (OSA). It will also assess the Morning Aligner as a supporting tool to maintain jaw alignment and comfort.

   In addition to following patients prospectively over three years, this study will also analyze and compare pre-existing clinical data from other patients who have used different nylon-based mandibular advancement devices. This approach will allow us to assess relative performance in terms of treatment outcomes, comfort, and long-term adherence.
2. Hypothesis The OrthoApnea NOA, used with the Morning Aligner, will reduce the Apnea-Hypopnea Index (AHI) by at least 50%, with a goal of bringing AHI to fewer than 5 events per hour in many patients.

   Compared to other nylon-based dental appliances, the NOA will show:

   Better long-term efficacy

   Longer retention time (device durability)

   Higher adherence to treatment

   Improved patient comfort and satisfaction
3. Justification Dental sleep appliances are a valuable alternative for patients who cannot tolerate continuous positive airway pressure (CPAP) therapy. The OrthoApnea NOA is a custom-made, modern appliance designed for maximum comfort, adjustability, and effectiveness. Including the Morning Aligner in the treatment may enhance comfort and prevent bite changes.

   There is currently limited long-term real-world data comparing this device with other nylon-based appliances. This study aims to fill that gap by evaluating both new patients and historical patient data, providing robust evidence to support treatment decisions.
4. Objectives Primary Objective To evaluate whether the OrthoApnea NOA reduces AHI by ≥50%, with a goal of achieving <5 events per hour.

   Secondary Objectives

   Measure improvements in:

   AHI (Apnea-Hypopnea Index)

   CT90 (percentage of time with oxygen saturation below 90%)

   BMI (body mass index)

   Epworth Sleepiness Scale (ESS) scores

   Device retention/durability

   Jaw alignment and dental comfort

   Patient adherence and satisfaction
5. Study Design and Methods Design Quasi-experimental, comparative longitudinal study

   Two groups:

   Prospective cohort using the OrthoApnea NOA + Morning Aligner

   Retrospective cohort of patients treated with other nylon-based oral appliances (existing clinic data)

   Sample

   Total Sample Size: 250

   Intervention Sample Size: 100 patients in the prospective NOA group

   Historical Comparison Group: 100-150 matched patients from prior records

   Sample Size and Power Calculation

   Calculated using the Harvard Hedwig sample size calculator sing a 2 sided alpha of 0.05, power of 0.9 with a standard deviation of 10 and a difference in means of 5 and a dropout rate of approximately 20% for the prospective group
6. Data Collection and Follow-up

   Prospective Group (OrthoApnea NOA + Morning Aligner):

   Sleep studies at baseline, 6, 12, 18, 24, and 36 months

   CT90, BMI, ESS, and dental/jaw evaluations

   Patient questionnaires on comfort, satisfaction, and adherence

   Device assessments for wear and retention

   Retrospective Group (Other nylon appliances):

   Extract AHI, CT90, BMI, ESS, and device durability from patient records

   Match based on age, gender, OSA severity, and BMI
7. Data Analysis Plan Primary Analysis

Compare changes in AHI from baseline to follow-up between the NOA group and retrospective nylon appliance group using:

Independent t-tests or ANCOVA for continuous variables (adjusting for baseline values)

Chi-square tests for categorical outcomes (e.g., proportion of patients achieving AHI < 5)

Secondary Analyses Longitudinal trends in AHI, CT90, ESS, and BMI using mixed-effects models

Analysis of device durability and patient adherence using survival analysis or time-to-event methods

Evaluate correlations between adherence, comfort, and clinical improvement

Subgroup analysis by OSA severity (mild, moderate, severe)

Data Matching and Control

Retrospective data will be matched to prospective participants based on:

Age Sex Baseline AHI category BMI Propensity score matching may be used for more accurate comparisons

This study combines real-world clinical data with a prospective follow-up to evaluate the long-term effectiveness of the OrthoApnea NOA appliance and its companion Morning Aligner. It will provide strong, comparative evidence of its performance against other nylon-based devices in terms of sleep improvement, patient comfort, and adherence-information that is critically needed for guiding future treatment recommendations in dental sleep medicine.

ELIGIBILITY:
Inclusion Criteria:

* Dxed OSA being treated with NOA appliance

Exclusion Criteria:

* no OSA Dx

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults with OSA
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-09-30 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
AHI | 3 years
  Disease Index

SECONDARY OUTCOMES:
Side Effects | 3 years
  Side Effects (changes to bite/occlusion, TMJ symptoms/myalgia)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No